CLINICAL TRIAL: NCT07130370
Title: Effectiveness of Mindfulness-informed Intervention for Diabetes-related Outcomes Among Individuals With Type 2 Diabetes
Brief Title: Mindfulness-informed Intervention for Improving Diabetes Outcomes in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Modern Languages (Other)
Responsible Party: Principal Investigator, Faiza Batool, Lecturer, National University of Modern Languages
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NationalUModernLanguages
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes (T2DM)
Keywords: Mindfulness, Acceptance and commitment therapy, diabetes distress, psychological flexibility, diabetes self-care practice; Mindfulness; Acceptance and commitment Therapy; Type 2 Diabetes; Diabetes Distress; Diabetes Self-care Practice; Psychological Flexibility
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-informed Acceptance and commitment Therapy (Experimental): In this arm, culturally adapted acceptance and commitment therapy will be utilized to improve diabetes outcomes among individuals with type 2 diabetes
  Interventions: Behavioral: Acceptance and commitment therapy
- Waitlist Control Group (No Intervention): This group would be receiving routine diabetes treatment by primary health care provider (Treatment as usual).

INTERVENTIONS:
Behavioral: Acceptance and commitment therapy — Acceptance and Commitment Therapy (ACT) is a mindfulness-informed behavioral intervention that helps individuals accept difficult thoughts and feelings, clarify personal values, and commit to meaningful actions. It aims to improve psychological flexibility, enabling healthier coping with life's challenges.
  Arms: Mindfulness-informed Acceptance and commitment Therapy

SUMMARY:
The goal of this clinical trial is to learn if Acceptance and Commitment Therapy (ACT), a mindfulness-based psychological approach, can improve health and emotional well-being in adults with type 2 diabetes.

The main questions it aims to answer are:

Can ACT reduce diabetes-related distress?

Can ACT improve self-care behaviors?

Can ACT improve psychological flexibility?

Researchers will compare people who receive ACT to those in a waitlist control group to see if ACT has better effects on diabetes-related outcomes.

Participants will:

Attend ACT sessions tailored for people with type 2 diabetes

Complete questionnaires about their health, mood, and self-care.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) is a chronic metabolic disorder that requires ongoing medical care and self-management to prevent acute complications and reduce the risk of long-term complications. In addition to physical health challenges, many individuals with T2DM experience high levels of diabetes distress (DD), decreased self-efficacy, and difficulties in sustaining recommended lifestyle behaviors. Psychological interventions targeting these factors may enhance both mental and physical health outcomes.

Acceptance and Commitment Therapy (ACT), a third-wave behavioral therapy, emphasizes mindfulness, acceptance of internal experiences, and commitment to value-driven action. ACT aims to increase psychological flexibility - the ability to remain engaged in meaningful activities even when faced with difficult thoughts, emotions, or physical sensations. Although ACT has shown efficacy for various chronic illnesses, there is limited evidence from randomized controlled trials (RCTs) in Pakistan, and none to date for T2DM populations in this setting.

This randomized controlled trial will evaluate the effectiveness of a culturally adapted, group-based ACT program for adults diagnosed with T2DM. The primary objectives are:

To determine whether ACT reduces diabetes distress.

To assess whether ACT improve diabetes self-care behaviors, diabetes distress, diabetes self efficacy, psychological flexibility, self-compassion, coping and perceived social support

Study Design:

Type: Interventional, randomized, parallel-assignment clinical trial.

Participants: Adults (≥18 years) with a diagnosis of T2DM for at least 1 year, able to attend group sessions, moderate to high diabetes distress and providing informed consent.

Sample Size: 50 participants

Arms:

ACT Intervention Group: Participants will attend weekly, 60min group sessions for 6 weeks. The program will integrate mindfulness practices, acceptance-based coping strategies, and value clarification tailored for individuals with T2DM in Pakistan.

Waitlist Control Group: Participants will receive standard medical care during the study period and will be offered the ACT program after study completion.

Outcome Measures:

Primary Outcome: Change in diabetes distress, diabetes self-care practices and psychological flexibility from baseline to post-intervention.

Secondary Outcomes: changes in diabetes self-efficacy, self-compassion, perceived social support and coping.

Data Collection Timeline:

T1: Baseline assessment (questionnaires).

T2: Immediately post-intervention.

Significance:

This study will be the first RCT in Pakistan to examine the impact of ACT on diabetes-related outcomes in adults with T2DM. Findings will contribute to the global evidence base on ACT for chronic illness management and provide culturally relevant recommendations for integrating psychological care into diabetes management in low- and middle-income countries.

ELIGIBILITY:
Inclusion Criteria:

* having diagnosis of type 2 diabetes at least since one year and having moderate to high diabetes distress.

Exclusion Criteria:

* Psychosis, Dementia, Terminal Renal failure or other life threatening condition

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Diabetes Distress Assessment Scale | Before intervention and after six weeks of intervention
  It is a five point liker scale where "5" means there is a "serious problem" and 1 means "there is a not a problem". high score indicates greater level of diabetes distress.
Summary of Diabetes-Self-care activity | Before intervention and after six weeks of intervention
  It is 15 item scale to measure diabetes self-care practices. It is based on number of activities being performed the last week. Therefore response scale is from 0 till 7. where "0" means this particular self care activity has not been performed in the last week and "7" means it has been performed every day. Higher the score, higher the number of diabetes self-care practices performed last week. These include diet, blood glucose testing, Exercise, Foot care and Medications.

SECONDARY OUTCOMES:
Brief Coping Inventory | Before intervention and after six weeks of intervention
  It is translated version of BRIEF Cope Scale (Brief Coping Inventory) in Urdu. It is a four point liker scale from 0-4. Where higher score indicates greater level of particular coping strategy is used by the individual. The subscales include emotion-focused coping, problem-focused coping and avoidance coping.

CONTACTS AND LOCATIONS:
Overall Officials: Anila Sadaf, PhD, Study Director — National University of Modern Languages, Islamabad
Locations (1):
- University Counseling Centre, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No
It will be shared upon request.

REFERENCES:
- [Background] Fisher L, Polonsky WH, Perez-Nieves M, Desai U, Strycker L, Hessler D. A new perspective on diabetes distress using the type 2 diabetes distress assessment system (T2-DDAS): Prevalence and change over time. J Diabetes Complications. 2022 Aug;36(8):108256. doi: 10.1016/j.jdiacomp.2022.108256. Epub 2022 Jul 5. PMID 35810147
- See also: Publication of article on systemic review — https://pakjmcr.com/index.php/1/article/view/67
- Available data/document: Informed Consent Form: fabatool@numl.edu.pk — https://pakjmcr.com/index.php/1/article/view/67 — It is not applicable at this time.